CLINICAL TRIAL: NCT07401433
Title: Efficacy Of Levetiracetam in the Treatment of Neonatal Seizures Presenting at Tertiary Care Hospital.
Brief Title: Levetiracetam Versus Phenobarbitone for the Treatment of Neonatal Seizures in a Tertiary Care Hospital.
Acronym: LEV-NEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hayat Abad Medical Complex, Peshawar (Other Government)
Collaborators: Gomal Medical College (Other)
Responsible Party: Principal Investigator, Gohar Ali, Trainee Registrar, Hayat Abad Medical Complex, Peshawar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DHQ-DIK-IREB NO. 4806
Record Dates: First submitted 2026-01-17; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neonatal Seizures
Keywords: Neonatal seizures; Levetiracetam; Phenobarbitone; Antiepileptic drugs; Neonatal intensive care
MeSH Terms: interventions — Levetiracetam; Phenobarbital

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel treatment groups: intravenous levetiracetam or phenobarbitone-based therapy, with no crossover between groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, treating clinicians, investigators, and outcome assessors were blinded to treatment allocation. Randomization was performed using sealed opaque envelopes to maintain allocation concealment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levitiracetam Group (Experimental): Neonates presenting with clinically diagnosed seizures will receive intravenous levetiracetam as the first-line anticonvulsant. Initial dose 20 mg/kg IV, followed by 20 mg/kg IV after 12 hours if seizures persist. Maintenance dose will be 10 mg/kg IV/PO twice daily as per hospital protocol. Seizure control and side effects will be monitored.
  Interventions: Drug: Levetiracetam
- Phenobarbitone Group (Active Comparator): Neonates with clinically diagnosed seizures received intravenous phenobarbitone as the first-line anticonvulsant with a loading dose of 20 mg/kg followed by maintenance dosing of 3-5 mg/kg/day. In cases of persistent seizures, phenytoin was added according to standard dosing protocols. Seizure response and adverse effects were monitored.
  Interventions: Drug: Phenobarbital Sodium Injection

INTERVENTIONS:
Drug: Levetiracetam — Neonates with clinically diagnosed seizures received intravenous levetiracetam as the first-line anticonvulsant. Levetiracetam was administered at a rate of 1 mg/kg/min followed by a loading dose of 20 mg/kg diluted in normal saline. Maintenance therapy of 20 mg/kg/day was continued after seizure control. Seizure response and adverse effects were monitored.
  Arms: Levitiracetam Group
Drug: Phenobarbital Sodium Injection — Phenobarbitone will be administered intravenously as the first-line anticonvulsant for neonatal seizures. Initial loading dose 20 mg/kg IV. If seizures persist after 20 minutes, a second dose of 10 mg/kg IV will be given. Maintenance dose of 5 mg/kg IV/PO once daily will be continued until seizure control is achieved or until discharge. Seizure response and adverse effects will be monitored.
  Arms: Phenobarbitone Group

SUMMARY:
Neonatal seizures are a common neurological emergency in newborn babies and can lead to serious brain injury if not treated promptly. Phenobarbitone is commonly used as first-line treatment, but it is associated with delayed seizure control and adverse effects such as sedation and poor feeding.

This study was conducted to compare the effectiveness and safety of levetiracetam with conventional antiepileptic drugs (phenobarbitone with or without phenytoin) in the treatment of neonatal seizures.

In this randomized controlled trial, newborns aged 0 to 28 days diagnosed with seizures were randomly assigned to receive either intravenous levetiracetam or phenobarbitone-based therapy. The main outcomes assessed were seizure control within 40 minutes, seizure freedom at 24 and 48 hours, recurrence of seizures, time taken to control seizures, adverse effects, and mortality.

The results of this study aim to provide evidence on whether levetiracetam is a safer and more effective alternative for managing neonatal seizures in a tertiary care hospital setting.

DETAILED DESCRIPTION:
This study is a prospective, double-blinded, randomized controlled parallel-group trial conducted in the Neonatal Intensive Care Unit of the Department of Pediatrics, MTI District Head Quarter Hospital, Dera Ismail Khan. The study was carried out over a period of one year after approval from the Institutional Research and Ethics Board.

A total of 260 neonates aged 0 to 28 days with clinically diagnosed neonatal seizures were enrolled after obtaining written informed consent from parents or legal guardians. Neonates who were already receiving antiepileptic drugs or had congenital cardiac or renal diseases were excluded. Participants were randomly allocated into two equal groups using a table of random numbers with allocation concealment through sequentially numbered sealed opaque envelopes.

Group A received intravenous levetiracetam administered at a rate of 1 mg/kg/min, followed by a loading dose of 20 mg/kg diluted in normal saline. Maintenance therapy of 20 mg/kg/day was continued after seizure control. Group B received phenobarbitone as first-line therapy with a loading dose of 20 mg/kg followed by maintenance dosing. In cases of persistent seizures, phenytoin was added according to standard dosing protocols. No crossover between groups occurred.

The primary outcome was seizure cessation within 40 minutes of drug administration. Secondary outcomes included seizure freedom at 24 and 48 hours, recurrence of seizures, mean time to seizure control, adverse effects such as sedation, respiratory suppression, hypotension, and mortality. All patients were monitored in the neonatal intensive care unit for five days and followed for up to 14 weeks after discharge.

Data were analyzed using SPSS software. Outcomes were compared between groups to evaluate the efficacy and safety of levetiracetam compared with phenobarbitone-based therapy in the management of neonatal seizures.

ELIGIBILITY:
Inclusion Criteria:

* Neonates (0-28 days old) with clinically diagnosed seizures.
* Both term and preterm neonates.
* Admitted to the neonatal intensive care unit (NICU) or pediatric ward.
* Written informed consent obtained from parents or legal guardians.

Exclusion Criteria:

* Neonates with major congenital anomalies or genetic syndromes.
* Neonates with severe renal or hepatic impairment.
* Neonates with metabolic disorders requiring specific treatment (e.g., hypoglycemia, hypocalcemia) unless seizures persist after correction.
* Neonates already receiving anticonvulsant therapy prior to admission.
* Neonates with confirmed meningitis or central nervous system infections requiring specific management (unless seizures persist after appropriate treatment).
* Neonates with life-threatening conditions where study treatment cannot be safely administered.
* Parents or legal guardians refusing consent.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Seizure Cessation Within 40 Minutes | Immediately after first-line drug administration (within 40 minutes)
  Proportion of neonates with clinically diagnosed seizures whose seizures stopped completely within 40 minutes after administration of the first-line anticonvulsant.

SECONDARY OUTCOMES:
Time to Seizure Cessation | From first-line drug administration to seizure cessation (up to 40 minutes)
  Time duration from administration of the first dose to complete cessation of seizures.
Need for Second-Line Anticonvulsant | Immediately after first-line treatment failure (within 40 minutes of initial drug administration)
  Proportion of neonates requiring second-line anticonvulsant therapy due to failure of initial treatment.
Seizure Recurrence During Hospital Stay | From initial seizure control through 7 days of hospitalization
  Number of neonates who develop recurrent seizures after initial control during the hospital stay.
Incidence of Adverse Drug Reactions | From first drug administration through the first 5 days of hospitalization
  Incidence of adverse effects (e.g., sedation, hypotension, respiratory depression, rash, feeding intolerance) associated with levetiracetam or phenobarbitone.
Mortality | From enrollment through assessment at discharge, 28 days and 90days
  Number of deaths occurring during hospital stay among neonates treated with levetiracetam or phenobarbitone.

CONTACTS AND LOCATIONS:
Locations (1):
- Gomal Medical College, Dera Ismāīl Khān, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study is conducted at a single tertiary care hospital with limited resources, and the dataset contains sensitive clinical information of neonates. Data confidentiality and privacy of participants will be maintained in accordance with institutional ethical guidelines. Only aggregate data and study results will be published. De-identified data may be shared upon reasonable request and approval from the institutional ethics committee.

REFERENCES:
- [Result] İşgüder R, Güzel O, Ağın H, Yılmaz Ü, Akarcan SE, Çelik T, et al. - Efficacy and Safety of IV Levetiracetam in Children With Acute Repetitive Seizures. Pediatric Neurology. 2014 Nov;51(5):688-95.
- [Result] Khan O, Cipriani C, Wright C, Crisp E, Kirmani B - Role of intravenous levetiracetam for acute seizure management in preterm neonates. Pediatr Neurol. 2013 Nov;49(5):340-3.
- [Result] Sourbron J, Chan H, Heijden EAW van der, Klarenbeek P, Wijnen BFM, Haan GJ de, et al. - Review on the relevance of therapeutic drug monitoring of levetiracetam. Seizure - European Journal of Epilepsy. 2018 Nov;62:131-5.
- [Result] Efficacy of levetiracetam as the first line antiepileptic drug in neonatal seizures (ResearchGate PDF).
- [Result] Sharpe C, Reiner GE, Davis SL, Nespeca M, Gold JJ, Rasmussen M, et al. - Levetiracetam Versus Phenobarbital for Neonatal Seizures: A Randomized Controlled Trial. Pediatrics. 2020 Jun;145(6):e20193182.
- [Result] McHugh DC, Lancaster S, Manganas LN - A Systematic Review of the Efficacy of Levetiracetam in Neonatal Seizures. Neuropediatrics. 2018 Feb;49(1):12-7.
- [Result] Weldegerima K, Gebremariam DS, Haftu H, Berhe G, Hadgu A, Mohammedamin MM - Neonatal Seizure Pattern, Outcome, and its Predictors Among Neonates Admitted to NICU of Ayder Comprehensive Specialized Hospital, Mekelle, Tigray, Ethiopia. Int J Gen Med. 2023;16:4343-55.
- [Result] Kaminiow K, Kozak S, Paprocka J. Neonatal Seizures Revisited. Children (Basel). 2021 Feb 18;8(2):155. doi: 10.3390/children8020155. PMID 33670692
- [Result] Ramantani G, Schmitt B, Plecko B, Pressler RM, Wohlrab G, Klebermass-Schrehof K, Hagmann C, Pisani F, Boylan GB. Neonatal Seizures-Are We there Yet? Neuropediatrics. 2019 Oct;50(5):280-293. doi: 10.1055/s-0039-1693149. Epub 2019 Jul 24. PMID 31340400

DOCUMENTS (2):
  • Study Protocol (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT07401433/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT07401433/SAP_001.pdf